CLINICAL TRIAL: NCT03650023
Title: A Crossover Trial of Chitosan Oligosaccharide (GO2KA1) on Post Prandial Glucose Control in Subjects With Normal Blood Glucose, Impaired Fasting Glucose and Impaired Glucose Tolerance
Brief Title: A Crossover Trial of Chitosan Oligosaccharide on Post Prandial Glucose Control in Subjects With Normal, IFG and IGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, PI, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCK_OFTT
Record Dates: First submitted 2018-08-26; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Normal; Impaired Fasting Glucose; Impaired Glucose Tolerance
Keywords: Chitosan Oligosaccharide; diabetes mellitus; blood glucose; fasting blood sugar; normal blood glucose; impaired fasting glucose; Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — GO2KA1; Egg White

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitosan Oligosaccharide (GO2KA1) (Experimental): Chitosan Oligosaccharide (GO2KA1) capsule was provided to the study participants. The Chitosan Oligosaccharide (GO2KA1) capsule was consumed within 15 min, and then 2-h oral sucrose tolerance test was conducted. The Chitosan Oligosaccharide (GO2KA1) one capsule had Chitosan Oligosaccharide 250mg.
  Interventions: Dietary Supplement: Chitosan Oligosaccharide (GO2KA1)
- White egg (Placebo Comparator): White egg capsule was provided to the study participants. The White egg capsule was consumed within 15 min, and then 2-h oral sucrose tolerance test was conducted. The Chitosan Oligosaccharide (GO2KA1) one capsule had White egg 250mg.
  Interventions: Dietary Supplement: White egg

INTERVENTIONS:
Dietary Supplement: Chitosan Oligosaccharide (GO2KA1) — Chitosan Oligosaccharide (GO2KA1) capsule was consumed within 15 min, and then 2-h oral sucrose tolerance test was conducted.
  Arms: Chitosan Oligosaccharide (GO2KA1)
Dietary Supplement: White egg — White egg capsule was consumed within 15 min, and then 2-h oral sucrose tolerance test was conducted.
  Arms: White egg

SUMMARY:
It is well known that Chitosan oligosaccharide is low molecular weight and water soluble and chitosan oligosaccharide has been shown to reduce blood cholesterol and blood pressure, increase immunity, and enhance antitumor properties. the effect of chitosan oligosaccharide (GO2KA1) supplementation on glucose control in subjects with normal blood glucose, impaired fasting glucose and impaired glucose tolerance.

DETAILED DESCRIPTION:
A randomized, double-blinded, controlled, cross-over trial was conducted to verify the effects of chitosan oligosaccharide (GO2KA1). forty healthy male and female subjects aged 20-75 years with normal blood glucose, impaired fasting glucose and impaired glucose tolerance were recruited. The subjects visited the research site twice over with a seven-day interval after an overnight fast at least 12 hr. On the screening visit, the participants were the 2-hr oral glucose tolerance test (OGTT) was conducted. And they were separated normal blood glucose, impaired fasting glucose and impaired glucose tolerance. On the first visit, the participants were randomly assigned to consume a test or placebo product [test product: chitosan oligosaccharide powder 500mg (GO2KA1); placebo product: white egg powder 500mg] and ingested the assigned product. On the second visit, the participants consumed the other product that they did not eat on the first visit. On both visit day, the 2-hr oral sucrose tolerance test (OSTT) was conducted and started at 8:00 in the morning; venous blood samples were collected before (0 hr) and after ingestion (0.5, 1 and 2 hr) of the products.

ELIGIBILITY:
Inclusion Criteria:

* Normal Blood Glucose (fasting blood sugar below 100mg/dl, two hours after meals below 140mg/dl)
* Impaired Fasting Glucose (fasting blood sugar 100-125mg/dl)
* Impaired Glucose Tolerance (two hours after meals 140-199mg/dl)

Exclusion Criteria:

* history/presence of diabetes mellitus (including oral hypoglycaemic agent and insulin)
* history of serious hypoglycemia
* history of serious cardiovascular, cerebrovascular disease, pulmonary, gastrointestinal, hepatic, renal and/or haematological disease
* uncontrolled blood pressure (blood pressure level more than 140/90mmHg)
* history/presence of alcoholism, drug addiction, etc.
* taking a regulation of blood glucose medications within 1 month before study
* participation other intervention studies within 1 months before study
* history of diagnosed with cancer, cancer surgery and hospitalization
* women who are pregnant or desire to become pregnant during the study period
* having any other medical condition which, in the opinion of the investigator, could interfere with participation in the study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 2 hours
  Glucose level differences during the 2-hr oral sucrose tolerance test between White egg and chitosan oligosaccharide (GO2KA1) intak

SECONDARY OUTCOMES:
The areas under the curve (AUC) of glucose | 1 day of second visit (after finishing cross-over trial)
  Glucose AUC differences between White egg and chitosan oligosaccharide (GO2KA1) intake

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

REFERENCES:
- [Derived] Jeong S, Min Cho J, Kwon YI, Kim SC, Yeob Shin D, Ho Lee J. Chitosan oligosaccharide (GO2KA1) improves postprandial glycemic response in subjects with impaired glucose tolerance and impaired fasting glucose and in healthy subjects: a crossover, randomized controlled trial. Nutr Diabetes. 2019 Nov 4;9(1):31. doi: 10.1038/s41387-019-0099-4. PMID 31685797